CLINICAL TRIAL: NCT06685471
Title: Simulation-Based Training Program Effect on Pediatric Nurses' Knowledge and Performance Regarding Heel-Prick During Newborn Blood Screening Test
Brief Title: Simulation-Based Training Program Effect on Pediatric Nurses Regarding Heel-Prick Screening Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abeer Abd Elwahed Almowafy (Other)
Responsible Party: Sponsor-Investigator, Abeer Abd Elwahed Almowafy, Clinical Professor, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: UB-RELOC H-06-BH-089)/ 1204.24
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Aspiration of Blood in Newborn

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation-Based Training Program Effect on Pediatric Nurses' Knowledge and Performance (Experimental): Simulation-Based Training Program
  Interventions: Diagnostic Test: Screeing test
- traditional method (No Intervention): traditional method program

INTERVENTIONS:
Diagnostic Test: Screeing test — Simulation-Based Training Program Effect on Pediatric Nurses' Knowledge and Performance Regarding Heel-Prick during Newborn Blood Screening Test
  Arms: Simulation-Based Training Program Effect on Pediatric Nurses' Knowledge and Performance

SUMMARY:
This study aimed to assess the impact of simulation-based training on pediatric nurses' knowledge and performance regarding the heel-prick technique used during newborn blood screening tests in select hospitals in Saudi Arabia and Egypt. This study utilized an experimental pre-test and post-test design. The G*Power Program® Version 3.1.9.4 was employed to determine the necessary sample size to fulfill the study's objectives. The sample consisted of 50 nurses recruited from the Maternity & Children Hospital Bisha, Al-Namas General Hospital in the Kingdom of Saudi Arabia, and Pediatric Assiut University Hospital in Egypt. The current study's findings indicate that, following simulation-based training, pediatric nurses significantly improved their heel-prick knowledge and performance during the newborn blood screening test. This study provides strong evidence that the simulation-based training program improved nurses' knowledge and performance, and we advise all pediatric healthcare practitioners, physicians, and nurses employed in hospitals and healthcare facilities to undergo advanced simulation-based training. Nursing managers can target public hospitals with low scores by putting systematic methods into place to improve nurses' performance and knowledge in simulation-based training.

DETAILED DESCRIPTION:
One of the best ways to impart important skills to trainees is through simulation-based training which is more reliable than the conventional method of doing clinical examinations. It is used in pediatric nursing training to allow nurses to practice and improve their clinical and conversational skills during an actual child encounter. A heel-prick is a complex psychomotor task that requires skill and knowledge on the part of the pediatric nurse who is performing the procedure while applying for the National Newborn Screening Program.

ELIGIBILITY:
Inclusion Criteria:The study's inclusion criteria encompassed nurses, regardless of their age, gender, education, experience, part-time status, or administrative responsibilities, who gave their consent to participate. Pediatric nurses in experimental and control groups had recently graduated, worked for less than 6 months, and did not have any training program by simulation-based training for using the Newborn Blood Spot Test Simulator regarding heel-pricks during newborn blood screening tests.

-

Exclusion Criteria:The exclusion criteria included nursing experience for more than six months, as well as non-consenting participants.

-

Ages: 25 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
• pediatric nurses' knowledge in newborn blood screening tests compared to traditional training methods | 8 week
  • Simulation-based training will increase the pediatric nurses' knowledge in newborn blood screening tests compared to traditional training methods.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Almowafy, Principal Investigator — Al-Azhar University
Locations (1):
- Abeer, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asiri A, Almowafy AA, Moursy SM, Abd-Elhay HA, Ahmed SAK, Abdelrahem AS, Seif MTA, Ahmed FA. Simulation-based training program effect on pediatric nurses' knowledge and performance regarding heel-prick during newborn blood screening test. BMC Nurs. 2025 Jan 29;24(1):110. doi: 10.1186/s12912-024-02657-7. PMID 39881378